CLINICAL TRIAL: NCT01397578
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter, Phase II Study to Evaluate the Impact of MABT5102A on Brain Amyloid Load and Related Biomarkers in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Study to Evaluate the Impact of MABT5102A on Brain Amyloid Load and Related Biomarkers in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABE4955g; GN00762 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Part 1: Subcutaneous cohort exp (Experimental)
  Interventions: Drug: MABT5102A
- Part 2: Intravenous cohort exp (Experimental)
  Interventions: Drug: MABT5102A
- Part 1: Subcutaneous cohort (Placebo Comparator): Repeating subcutaneous injection
  Interventions: Drug: placebo
- Part 2: Intravenous cohort (Placebo Comparator): Repeating intravenous injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MABT5102A — Repeating subcutaneous injection
  Arms: Part 1: Subcutaneous cohort exp
Drug: MABT5102A — Repeating intravenous infusion
  Arms: Part 2: Intravenous cohort exp
Drug: placebo — Repeating subcutaneous injection
  Arms: Part 1: Subcutaneous cohort
Drug: placebo — Repeating intravenous infusion
  Arms: Part 2: Intravenous cohort

SUMMARY:
This is a Phase II, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the effects of MABT5102A on brain amyloid burden (as assessed by amyloid PET imaging) and other biomarkers in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorder Association (NINCDS-ADRDA) criteria
* Mini-Mental State Examination (MMSE) score of 18-26 points at screening
* Geriatric Depression Scale (GDS-15) score of < 6
* Completion of 6 years of education (or good work history consistent with exclusion of mental retardation or other pervasive developmental disorders)
* For patients currently receiving treatment with approved AD treatments (AChE inhibitors or memantine): Treatment initiated and continued for at least the last 3 months prior to randomization, at a stable dose for at least the last 2 months prior to randomization

Exclusion Criteria:

* Severe or unstable medical condition that, in the opinion of the investigator or Sponsor, would interfere with the patient's ability to complete the study assessments or would require the equivalent of institutional or hospital care
* History or presence of clinically evident vascular disease potentially affecting the brain (e.g., stroke, clinically significant carotid or vertebral stenosis or plaque, aortic aneurysm, intracranial aneurysm, cerebral hemorrhage, arteriovenous malformation)
* History of severe, clinically significant (persistent neurologic deficit or structural brain damage) central nervous system trauma (e.g., cerebral contusion)
* Hospitalization within 4 weeks prior to screening
* Previous treatment with MABT5102A or any other therapeutic that targets Abeta
* Treatment with any biologic therapy within 5 half-lives or 3 months prior to screening, whichever is longer, with the exception of routinely recommended vaccinations, which are allowed

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-08-31 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Change in brain amyloid load as assessed by amyloid PET imaging | Baseline to Week 69

SECONDARY OUTCOMES:
Changes in cerebrospinal fluid (CSF) biomarkers relevant to Alzheimer's disease | Baseline to Week 69
Change in brain metabolism as assessed by 18F-fluorodeoxyglucose positron emission tomography (FDG PET) imaging | Baseline to Week 69
Change in Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS Cog) score | Baseline to Week 73

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paul, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (29):
- United States (22):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - NNS Clinical Research LLC, Tucson, Arizona
  - Margolin Brain Institute, Fresno, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Pacific Neuroscience Med Grp, Oxnard, California
  - Stanford Univ Medical Center, Palo Alto, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Internal Med Assoc of Lee Cty, Fort Myers, Florida
  - Neuropsychiatric Research; Center of Southwest Florida, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - Compass Research, Orlando, Florida
  - Dekalb Neurology Associates, Decatur, Georgia
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Litwin Zucker Research Ctr.; Feinstein Inst. Med. Rsch., Manhasset, New York
  - Neurology & Neuroscience Ctr of Ohio, Toledo, Ohio
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
- France (3):
  - Hopital Central-CHU de Nancy; Pharmacie, Nancy
  - Hôpital Casselardit; Cons memoire, Toulouse
  - Clinique Psychiatrique Univ, Tours
- Spain (4):
  - Fundació ACE, BArcelon, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Mutua De Terrasa, Barcelona

REFERENCES:
- [Derived] Polhamus DG, Dolton MJ, Rogers JA, Honigberg L, Jin JY, Quartino A. Longitudinal Exposure-Response Modeling of Multiple Indicators of Alzheimer's Disease Progression. J Prev Alzheimers Dis. 2023;10(2):212-222. doi: 10.14283/jpad.2023.13. PMID 36946448
- [Derived] Yoshida K, Moein A, Bittner T, Ostrowitzki S, Lin H, Honigberg L, Jin JY, Quartino A. Pharmacokinetics and pharmacodynamic effect of crenezumab on plasma and cerebrospinal fluid beta-amyloid in patients with mild-to-moderate Alzheimer's disease. Alzheimers Res Ther. 2020 Jan 22;12(1):16. doi: 10.1186/s13195-020-0580-2. PMID 31969177
- [Derived] Salloway S, Honigberg LA, Cho W, Ward M, Friesenhahn M, Brunstein F, Quartino A, Clayton D, Mortensen D, Bittner T, Ho C, Rabe C, Schauer SP, Wildsmith KR, Fuji RN, Suliman S, Reiman EM, Chen K, Paul R. Amyloid positron emission tomography and cerebrospinal fluid results from a crenezumab anti-amyloid-beta antibody double-blind, placebo-controlled, randomized phase II study in mild-to-moderate Alzheimer's disease (BLAZE). Alzheimers Res Ther. 2018 Sep 19;10(1):96. doi: 10.1186/s13195-018-0424-5. PMID 30231896